CLINICAL TRIAL: NCT02751047
Title: Comparison Between Pressure Controlled Mechanical Ventilation and Manual Ventilation During Mask Ventilation for Induction of Anesthesia in Children
Brief Title: Manual Ventilation Versus Pressure Controlled Mechanical Ventilation in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, Jin-Tae Kim, Associated professor, Seoul National University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: H1602-094-741
Record Dates: First submitted 2016-04-22; First posted 2016-04-26 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2018-08

CONDITIONS: Ventilation
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Manual ventilation (Placebo Comparator): During anesthetic induction, facemask ventilation is performed by manual bagging, after setting adjustable pressure limiting (APL) valve at 13 cmH2O. During mask ventilation, gastric ultrasonography is continuously performed to detect gastric insufflation.
  Interventions: Other: manual ventilation
- Pressure controlled mechanical ventilation (Active Comparator): During anesthetic induction, facemask ventilation is performed with mechanical ventilator by pressure controlled mode, with inspiratory pressure of 13 cmH2O. During mask ventilation, gastric ultrasonography is continuously performed to detect gastric insufflation.
  Interventions: Other: Pressure controlled mechanical ventilation

INTERVENTIONS:
Other: manual ventilation — Facemask ventilation is performed by manual bagging with reservoir bag.
  Arms: Manual ventilation
Other: Pressure controlled mechanical ventilation — Facemask ventilation is performed with mechanical ventilator by pressure controlled mode.
  Arms: Pressure controlled mechanical ventilation

SUMMARY:
The investigator will compare the feasibility of manual ventilation and pressure-controlled mechanical ventilation during facemask ventilation in children. The hypothesis is that the incidence of gastric insufflation would be lower during pressure-controlled mechanical ventilation when compared to manual ventilation.

ELIGIBILITY:
Inclusion Criteria:

* Children with American Society of Anesthesiologist (ASA) physical status 1, 2
* Children with normal body mass index

Exclusion Criteria:

* Difficult airway management
* pulmonary disease
* upper respiratory infection
* risk of pulmonary aspiration
* intestinal obstruction or abdominal distension
* stroke history or moyamoya disease

Ages: 1 Month to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 154 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2016-11 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Incidence of gastric insufflation | During facemask ventilation (90 seconds)

SECONDARY OUTCOMES:
The number of patients with adequate tidal volume | During facemask ventilation (90 seconds)
  Tidal volume of 6 - 10 ml/kg

CONTACTS AND LOCATIONS:
Overall Officials: Jin-Tae Kim, PhD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided